CLINICAL TRIAL: NCT01154283
Title: A Randomized Crossover Study of Standard, Noninvasive Positive Pressure Ventilation (NIPPV) and Low Expiratory Pressure NIPPV in Amyotrophic Lateral Sclerosis (ALS) Patients
Brief Title: Study of Standard Noninvasive Positive Pressure Ventilation (NIPPV) and Low Expiratory Pressure NIPPV in ALS Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kirsten Gruis (Other)
Collaborators: ALS Association (Other)
Responsible Party: Sponsor-Investigator, Kirsten Gruis, Associate Professor, University of Michigan
Organization: University of Michigan (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: ALSA-9611
Record Dates: First submitted 2010-06-29; First posted 2010-06-30 (Estimated); Results first posted 2017-01-02 (Estimated); Last update posted 2017-01-02 (Estimated); Status verified 2016-11

CONDITIONS: Amyotrophic Lateral Sclerosis
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Bi-level, standard, NIPPV (Active Comparator): Standard NIPPV with both an inspiratory and expiratory positive airway pressure.
  Interventions: Device: Viasys® Healthcare, Pulmonetic Systems, lap-top ventilator (LTV machine)
- IPAP-only, NIPPV (Experimental): NIPPV with only inspiratory positive airway pressure, no expiratory positive airway pressure
  Interventions: Device: Viasys® Healthcare, Pulmonetic Systems, lap-top ventilator (LTV machine)

INTERVENTIONS:
Device: Viasys® Healthcare, Pulmonetic Systems, lap-top ventilator (LTV machine) — Noninvasive positive airway pressure ventilation

SUMMARY:
The purpose of the study is to test whether noninvasive positive pressure ventilation (NIPPV) without expiratory positive airway pressure (EPAP) (inspiratory positive airway pressure (IPAP)-only) will result in an increase in patient usage of NIPPV compared with standard, Bi-level NIPPV. Secondarily, the investigators will assess measures of dyspnea, quality of life, patient satisfaction, and side effects.

DETAILED DESCRIPTION:
Subjects will be randomized on a 1:1 basis to one of two groups differing in the sequence of NIPPV settings ((a) standard, Bi-level NIPPV followed by IPAP-only NIPPV or (b) IPAP-only NIPPV followed by standard, Bi-level, NIPPV). Subjects will then spend 6 weeks using the first NIPPV set-up before crossing over to the other NIPPV treatment for 6 weeks. At the beginning of the study, subjects will undergo approximately two hours of training and education by a respiratory therapist regarding proper use of the Viasys® Healthcare, Pulmonetic Systems, lap-top ventilators (LTV machine). They will be fitted with the appropriate NIPPV set-up. The patients will use the same mask interface with the study NIPPV machine that they were using with their NIPPV (bi-level positive airway pressure (BiPAP)) machine prior to study entry.

The patients will have two additional study visits after the consent/training session: one at the end of 6 weeks, after the first NIPPV treatment period (prior to crossing over to the second NIPPV treatment), and the second at the end of 12 weeks, after the second NIPPV treatment period.

NIPPV usage will be recorded as hours of use as measured objectively by the NIPPV machine hour meter. When the patient returns for his/her first study visit at the end of week six, the NIPPV machine hour meter will be recorded by the study investigator. By subtracting the hours recorded at the beginning of week two from the hours recorded at the end of week six, the NIPPV hours of usage for weeks two, three, four, five and six will be obtained. This same procedure will be repeated to record NIPPV hours of usage for the beginning of week eight and the end of week twelve to measure the hours of usage with the second NIPPV set-up for weeks eight, nine, ten, eleven and twelve. This allows study subjects one week to adjust to the new pressure settings of each treatment arm.

Dyspnea as measured by the transition dyspnea index (TDI), and quality of life as measured by the EuroQol Visual analogue scale(VAS) will be re-administered at both 6 and 12 week study visits by study personnel. Lastly, patient preference of NIPPV treatment will be subjectively assessed at the 12 week study visit on a Likert scale (definitely first treatment, probably first treatment, no preference, probably second treatment, definitely second treatment).

ELIGIBILITY:
Inclusion Criteria:

1. Age greater than 18 years
2. Definite or probable ALS by El Escorial criteria
3. Maximal inspiratory force < 60 cm/H2O or FVC <50% predicted (American College of Chest Physicians' criteria for initiating NIPPV)
4. Patients must have used NIPPV (typically administered as BiPAP) for at least 2 months
5. Currently using NIPPV ≥5 days a week with an EPAP = 4 cm H2O.

Exclusion Criteria:

1. Any medical condition that will interfere with participation
2. Inability to consent for him/herself
3. Known obstructive sleep apnea or obstructive pulmonary disease.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2008-01; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kirsten Gruis, MD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Bi-level, Standard, NIPPV Then IPAP-only NIPPV: Standard NIPPV with both an inspiratory and expiratory positive airway pressure then NIPPV with only inspiratory positive airway pressure (IPAP-only), no expiratory positive airway pressure
  Viasys® Healthcare, Pulmonetic Systems, lap-top ventilator (LTV machine): Noninvasive positive airway pressure ventilation (NIPPV)
- IPAP-only, NIPPV Then Bi-level, Standard NIPPV: NIPPV with only inspiratory positive airway pressure (IPAP-only), no expiratory positive airway pressure then Standard NIPPV with both an inspiratory and expiratory positive airway pressure
  Viasys® Healthcare, Pulmonetic Systems, lap-top ventilator (LTV machine): Noninvasive positive airway pressure ventilation (NIPPV)
Period: 0-6 Weeks
Arm/Group | Bi-level, Standard, NIPPV Then IPAP-only NIPPV | IPAP-only, NIPPV Then Bi-level, Standard NIPPV
Started | 14 | 14
Completed | 7 | 11
Not Completed | 7 | 3
Not completed — Withdrawal by Subject | 7 | 2
Not completed — Death | 0 | 1
Period: 7-12 Weeks
Arm/Group | Bi-level, Standard, NIPPV Then IPAP-only NIPPV | IPAP-only, NIPPV Then Bi-level, Standard NIPPV
Started | 7 | 11
Completed | 6 | 10
Not Completed | 1 | 1
Not completed — Death | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Bi-level, Standard, NIPPV Then IPAP-only NIPPV | IPAP-only, NIPPV Then Bi-level, Standard NIPPV | Total
Number analyzed (Participants) | 14 | 14 | 28
Age, Continuous [Mean (Full Range); unit: years] | 62 [48 to 78] | 59 [37 to 75] | 60 [37 to 78]
Gender [Count of Participants; unit: Participants]
  Female | 6 | 7 | 13
  Male | 8 | 7 | 15

OUTCOME MEASURES:

1. Primary Outcome: Hours of NIPPV Usage
Description: Patients experienced the first intervention period during weeks 1-6 and the second intervention period during weeks 7-12. Patients were given one week to learn how to use the NIPPV equipment at the beginning of each intervention period. Therefore, only the total NIPPV hours used during the last 5 weeks of each intervention period were collected and divided by the number of weeks to obtain the average, weekly hours of NIPPV usage assessed at 6 weeks (first intervention) and 12 weeks (second intervention) for each patient.
Time Frame: Assessed at 6 weeks (first intervention) and 12 weeks (second intervention)
Measure: Mean (Full Range); unit: hours
Arm/Group | Bi-level, Standard, NIPPV | IPAP-only, NIPPV
Number analyzed (Participants) | 17 | 17
hours | 49.94 [3.60 to 126.80] | 45.75 [0.00 to 159.20]

2. Secondary Outcome: Patient Preference (Likert Scale) "Definitely IPAP-only" "Probably IPAP-only" "Uncertain" "Probably Bi-level" "Definitely Bi-level"
Description: Patient Preference of NIPPV mode:
  definitely IPAP-only probably IPAP-only uncertain probably Bi-level definitely Bi-level Number of patients who chose definitely or probably are reported.
Time Frame: Assessed at 6 weeks (first intervention) and 12 weeks (second intervention)
Population: One patient died before completion of 12 weeks (second intervention) and could not have patient preference assessed.
Measure: Number; unit: participants
Arm/Group | Bi-level, Standard, NIPPV | IPAP-only, NIPPV
Number analyzed (Participants) | 16 | 16
participants | 2 | 12

3. Secondary Outcome: Transitional Dyspnea Index
Description: Transitional Dyspnea Index scores patient reported changes in difficulty breathing during each intervention period from -3 (major deterioration) to +3 (major improvement) in three categories: functional impairment, magnitude of task, and magnitude of effort. The total TDI score ranges from -9 to +9.
Time Frame: Assessed at 6 weeks (first intervention) and 12 weeks (second intervention)
Population: One patient died and unable to report dyspnea at end of 12 weeks. Two additional patients completed 12 weeks study but did not complete dyspnea assessments.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Bi-level, Standard, NIPPV | IPAP-only, NIPPV
Number analyzed (Participants) | 14 | 14
units on a scale | -3.14 (2.98) | -1.21 (2.72)

4. Secondary Outcome: EuroQol Visual Analogue Scale(VAS)
Description: Quality of life assessed with visual analogue scale. Where the patient is asked to place a mark on a piece of paper with a vertical, scale from 100 at the top to 0 at the bottom of the scale. Where the patient is informed that 100 represents his or her best imaginable health state and 0 is his or her worst imaginable health state.
Time Frame: Assessed at 6 weeks (first intervention) and 12 weeks (second intervention)
Population: One patient died and unable to report quality of life at end of 12 weeks. Two additional patients completed 12 weeks study but did not complete quality of life assessments.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Bi-level, Standard, NIPPV | IPAP-only, NIPPV
Number analyzed (Participants) | 14 | 14
units on a scale | 52.86 (25.32) | 62.79 (17.28)

ADVERSE EVENTS:
Time Frame: Collected during study intervention time frame of 12 weeks.
Groups:
- Bi-level, Standard, NIPPV: Standard NIPPV with both an inspiratory and expiratory positive airway pressure.
  Viasys® Healthcare, Pulmonetic Systems, lap-top ventilator (LTV machine): Noninvasive positive airway pressure ventilation (NIPPV)
- IPAP-only, NIPPV: NIPPV with only inspiratory positive airway pressure (IPAP-only), no expiratory positive airway pressure.
  Viasys® Healthcare, Pulmonetic Systems, lap-top ventilator (LTV machine): Noninvasive positive airway pressure ventilation (NIPPV)
Arm/Group | Bi-level, Standard, NIPPV | IPAP-only, NIPPV
Serious Adverse Events (participants affected / at risk) | 2/28 | 2/28
Other Adverse Events (participants affected / at risk) | 7/28 | 5/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bi-level, Standard, NIPPV (N=28) | IPAP-only, NIPPV (N=28)
Dysphagia (Gastrointestinal disorders) | 0 | 1 — Dysphagia led to hospitalization
Bronchial Disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Lower Respiratory Tract Infection (Infections and infestations) | 1 | 0
Urinary Tract Infection (Infections and infestations) | 0 | 1
Gastrointestinal motility and defaecation conditions (Gastrointestinal disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Bi-level, Standard, NIPPV (N=28) | IPAP-only, NIPPV (N=28)
Dysphagia (Gastrointestinal disorders) | 3 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 | 3
Cough Decreased (Respiratory, thoracic and mediastinal disorders) | 1 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No